CLINICAL TRIAL: NCT05462093
Title: Clinical Application of Annual Liver Multiscan and MRCP+ in Primary Sclerosing Cholangitis: the CATCH-IT Study
Brief Title: Clinical Application of Annual Liver Multiscan and MRCP+ in Primary Sclerosing Cholangitis
Acronym: CATCH-IT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Perspectum (Industry)
Responsible Party: Principal Investigator, C.Y. Ponsioen, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CATCH-IT
Record Dates: First submitted 2022-06-17; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Additional sequences with MRCP+ and LiverMultiscan (Other): PSC patients that undergo annual, standard care, MRI of the liver and MRCP will undergo additional Liver Multiscan sequences, taking approximately 15 minutes. After the MRI is performed, post-processing analysis named MRCP+ and LiverMultiscan will be performed without patient involvement.
  Interventions: Device: Liver Multiscan sequences; Device: Liver Multiscan analysis; Device: MRCP+

INTERVENTIONS:
Device: Liver Multiscan sequences — Additional Liver Multiscan sequences will be performed after the MRI liver with MRCP is performed, taking approximately 15 minutes.
Device: Liver Multiscan analysis — Post processing tool (Software) for determining the corrected T1 time after the additional LMS sequences at baseline are performed. This cT1 reflects the activity of inflammation/fibrosis of the liver. Patient involvement is not necessary during this procedure.
  Other Names: LMS
Device: MRCP+ — Post processing tool (Software) for quantifying MRCP images after the MRCP from follow up is performed. Patient involvement is not necessary during this procedure.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a chronic progressive biliary disease that affects approximately 1200 patients in the Netherlands and around 80,000 in the Western world. It is often accompanied by ulcerative colitis (UC) or Crohn's disease affecting the large bowel. The cause of PSC is unknown, there is no medical therapy available that has proven to halt disease progression and the median time until death or liver transplantation is 13-21 years.

Diagnosis is made by magnetic resonance cholangiography (MRC), or in the case of so called small duct disease by liver biopsy.

Due to the heterogeneous disease course and the relatively low clinical event rate of 5% per year it is difficult to predict prognosis of individual patients or to recommend any surveillance strategy for malignancies. Also, the lack of surrogate endpoints impedes performing clinical research. Recently, two new post-processing tools have been developed to characterize and quantify abnormalities in the biliary tree as well as excretory function captured by MRC. These tools called MRCP+ (quantitative magnetic resonance cholangiopancreatography +) and LiverMultiscan (LMS) hold the prospect of adequately depicting and quantifying lesions of the biliary tree as well as capturing functional derailment. However, several features must be tested before the utility of this tools in clinical patient care can be concluded. Therefore, the aim of this study is to investigate the utility of these novel techniques in monitoring disease activity by performing consecutive annual MRI's.

ELIGIBILITY:
Inclusion Criteria:

* Established PSC diagnosis according to the IPSCSG definitions
* Age ≥ 18
* Able to give informed consent

Exclusion Criteria:

* Post LTx
* Known allergy for MRI contrast agents, implants non-compatible with MRI or extreme claustrophobia causing discontinuation of MRI studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Delta of cT1 in patients with PSC during follow-up | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  The delta of cT1 (in ms), measured by LiverMultiscan, which will be assessed by performing paired t-tests.

SECONDARY OUTCOMES:
Assesment of th mean, median and range of cT1 and MRCP+ metrics in stable PSC patients | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52;
  Mean, median and range of cT1 and MRCP+ metrics in clinically and biochemically stable patients with PSC during the period of 1 year to establish general statistics as these are unknown at current writing
Variance of the delta of cT1 and MRCP+ metrics in stable patients | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Variance of the delta in cT1 and MRCP+ metrics from baseline to year 1 in clinically and biochemically stable patients
Difference in cT1 in patients with or without endoscopic intervention | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Difference in mean of cT1 values in patients who needed ERCP with treatment of dominant stricture(s) in the year following LMS measurement versus those who did not need an intervention
Variance in unstable patients | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Variance of the delta of cT1 and MRCP+ metrics in sequential scans in biochemically and/or clinically deteriorating patients.
Correlation of cT1 and MRCP+ metrics with fibroscan and MELD | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Correlation between cT1 and MRCP+ metrics with Fibroscan and MELD-score
Correlation of cT1 and MRCP+ metrics and development of dominant strictures | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Correlation between cT1 and MRCP+ metrics and development of dominant strictures
Correlation of cT1 and MRCP+ metrics and incidence of CCA | 1st MRI = baseline = week 0; 2nd MRI = year 1 = week 52; 3rd MRI = year 2 = week 104; 4th MRI = year 3 = week 156; 5th MRI = year 4 = week 208; 6th MRI = year 5 = week 260.
  Correlation between cT1 and MRCP+ metrics and incidence of CCA

CONTACTS AND LOCATIONS:
Overall Officials: Cyriel Ponsioen, Prof MD PhD, Principal Investigator — Gastroenterologist and hepatologist

IPD SHARING:
Plan to Share IPD: Yes
After publication, the following documentation can be requested by qualified research groups:
  - Study protocol, statistical analysis plan and the clinical study report can be provided if a proper request is submitted.
  IPD will contain decoded and only essential data for the objective of this study. Data that will be available for sharing purposes will only include decoded demographic data. Furthermore, MRCP+ data that underlies the results in the publication will be available for sharing, e.g. MRCP+ metrics
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Until 5 years after publication
Access Criteria: Data sharing can be requested by qualified research groups. Requests will be evaluated by the following method:
  The request is supposed to contain a clear objective and methodology. E.g., it must contain the objective to explore or validate the value of MRCP+ and LMS techniques. Furthermore, the study proposal could, for example, be a systematic review or meta-analysis.
  The request will be reviewed by a dedicated research team of the CATCH-IT-study. This research team contains the PI, PhD student, involved gastro-enterologist and radiologist and representative of Perspectum Ltd.
  If the request seems valid and the credibility of the requesting party is validated, data sharing agreement will be developed with the local research support team. To submit a request, contact t.e.middelburg@amsterdamumc.nl

REFERENCES:
- [Background] Lazaridis KN, LaRusso NF. Primary Sclerosing Cholangitis. N Engl J Med. 2016 Sep 22;375(12):1161-70. doi: 10.1056/NEJMra1506330. No abstract available. PMID 27653566
- [Background] Zheng HH, Jiang XL. Increased risk of colorectal neoplasia in patients with primary sclerosing cholangitis and inflammatory bowel disease: a meta-analysis of 16 observational studies. Eur J Gastroenterol Hepatol. 2016 Apr;28(4):383-90. doi: 10.1097/MEG.0000000000000576. PMID 26938805
- [Background] Barner-Rasmussen N, Pukkala E, Jussila A, Farkkila M. Epidemiology, risk of malignancy and patient survival in primary sclerosing cholangitis: a population-based study in Finland. Scand J Gastroenterol. 2020 Jan;55(1):74-81. doi: 10.1080/00365521.2019.1707277. Epub 2020 Jan 4. PMID 31902255
- [Background] Boonstra K, Weersma RK, van Erpecum KJ, Rauws EA, Spanier BW, Poen AC, van Nieuwkerk KM, Drenth JP, Witteman BJ, Tuynman HA, Naber AH, Kingma PJ, van Buuren HR, van Hoek B, Vleggaar FP, van Geloven N, Beuers U, Ponsioen CY; EpiPSCPBC Study Group. Population-based epidemiology, malignancy risk, and outcome of primary sclerosing cholangitis. Hepatology. 2013 Dec;58(6):2045-55. doi: 10.1002/hep.26565. Epub 2013 Oct 17. PMID 23775876
- [Background] Hirschfield GM, Karlsen TH, Lindor KD, Adams DH. Primary sclerosing cholangitis. Lancet. 2013 Nov 9;382(9904):1587-99. doi: 10.1016/S0140-6736(13)60096-3. Epub 2013 Jun 28. PMID 23810223
- [Background] Ponsioen CY, Chapman RW, Chazouilleres O, Hirschfield GM, Karlsen TH, Lohse AW, Pinzani M, Schrumpf E, Trauner M, Gores GJ. Surrogate endpoints for clinical trials in primary sclerosing cholangitis: Review and results from an International PSC Study Group consensus process. Hepatology. 2016 Apr;63(4):1357-67. doi: 10.1002/hep.28256. Epub 2015 Dec 23. PMID 26418478
- [Background] Ponsioen CY, Reitsma JB, Boberg KM, Aabakken L, Rauws EA, Schrumpf E. Validation of a cholangiographic prognostic model in primary sclerosing cholangitis. Endoscopy. 2010 Sep;42(9):742-7. doi: 10.1055/s-0030-1255527. Epub 2010 Jul 9. PMID 20623444
- [Background] Lindor KD, Kowdley KV, Harrison ME; American College of Gastroenterology. ACG Clinical Guideline: Primary Sclerosing Cholangitis. Am J Gastroenterol. 2015 May;110(5):646-59; quiz 660. doi: 10.1038/ajg.2015.112. Epub 2015 Apr 14. PMID 25869391
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases. J Hepatol. 2009 Aug;51(2):237-67. doi: 10.1016/j.jhep.2009.04.009. Epub 2009 Jun 6. No abstract available. PMID 19501929
- [Background] Berstad AE, Aabakken L, Smith HJ, Aasen S, Boberg KM, Schrumpf E. Diagnostic accuracy of magnetic resonance and endoscopic retrograde cholangiography in primary sclerosing cholangitis. Clin Gastroenterol Hepatol. 2006 Apr;4(4):514-20. doi: 10.1016/j.cgh.2005.10.007. PMID 16616358
- [Background] Dave M, Elmunzer BJ, Dwamena BA, Higgins PD. Primary sclerosing cholangitis: meta-analysis of diagnostic performance of MR cholangiopancreatography. Radiology. 2010 Aug;256(2):387-96. doi: 10.1148/radiol.10091953. PMID 20656832
- [Background] Chapman R, Fevery J, Kalloo A, Nagorney DM, Boberg KM, Shneider B, Gores GJ; American Association for the Study of Liver Diseases. Diagnosis and management of primary sclerosing cholangitis. Hepatology. 2010 Feb;51(2):660-78. doi: 10.1002/hep.23294. No abstract available. PMID 20101749
- [Background] Lunder AK, Hov JR, Borthne A, Gleditsch J, Johannesen G, Tveit K, Viktil E, Henriksen M, Hovde O, Huppertz-Hauss G, Hoie O, Hoivik ML, Monstad I, Solberg IC, Jahnsen J, Karlsen TH, Moum B, Vatn M, Negard A. Prevalence of Sclerosing Cholangitis Detected by Magnetic Resonance Cholangiography in Patients With Long-term Inflammatory Bowel Disease. Gastroenterology. 2016 Oct;151(4):660-669.e4. doi: 10.1053/j.gastro.2016.06.021. Epub 2016 Jun 21. PMID 27342213
- [Background] Zenouzi R, Welle CL, Venkatesh SK, Schramm C, Eaton JE. Magnetic Resonance Imaging in Primary Sclerosing Cholangitis-Current State and Future Directions. Semin Liver Dis. 2019 Jul;39(3):369-380. doi: 10.1055/s-0039-1687853. Epub 2019 Apr 30. PMID 31041791
- [Background] Goldfinger MH, Ridgway GR, Ferreira C, Langford CR, Cheng L, Kazimianec A, Borghetto A, Wright TG, Woodward G, Hassanali N, Nicholls RC, Simpson H, Waddell T, Vikal S, Mavar M, Rymell S, Wigley I, Jacobs J, Kelly M, Banerjee R, Brady JM. Quantitative MRCP Imaging: Accuracy, Repeatability, Reproducibility, and Cohort-Derived Normative Ranges. J Magn Reson Imaging. 2020 Sep;52(3):807-820. doi: 10.1002/jmri.27113. Epub 2020 Mar 8. PMID 32147892
- [Background] Tunnicliffe EM, Banerjee R, Pavlides M, Neubauer S, Robson MD. A model for hepatic fibrosis: the competing effects of cell loss and iron on shortened modified Look-Locker inversion recovery T1 (shMOLLI-T1 ) in the liver. J Magn Reson Imaging. 2017 Feb;45(2):450-462. doi: 10.1002/jmri.25392. Epub 2016 Jul 23. PMID 27448630
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Pavlides M, Banerjee R, Tunnicliffe EM, Kelly C, Collier J, Wang LM, Fleming KA, Cobbold JF, Robson MD, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging for the assessment of non-alcoholic fatty liver disease severity. Liver Int. 2017 Jul;37(7):1065-1073. doi: 10.1111/liv.13284. Epub 2017 May 30. PMID 27778429
- [Background] Bachtiar V, Kelly MD, Wilman HR, Jacobs J, Newbould R, Kelly CJ, Gyngell ML, Groves KE, McKay A, Herlihy AH, Fernandes CC, Halberstadt M, Maguire M, Jayaratne N, Linden S, Neubauer S, Banerjee R. Repeatability and reproducibility of multiparametric magnetic resonance imaging of the liver. PLoS One. 2019 Apr 10;14(4):e0214921. doi: 10.1371/journal.pone.0214921. eCollection 2019. PMID 30970039
- [Background] Pavlides M, Banerjee R, Sellwood J, Kelly CJ, Robson MD, Booth JC, Collier J, Neubauer S, Barnes E. Multiparametric magnetic resonance imaging predicts clinical outcomes in patients with chronic liver disease. J Hepatol. 2016 Feb;64(2):308-315. doi: 10.1016/j.jhep.2015.10.009. Epub 2015 Nov 10. PMID 26471505
- [Background] Bradley CR, Cox EF, Scott RA, James MW, Kaye P, Aithal GP, Francis ST, Guha IN. Multi-organ assessment of compensated cirrhosis patients using quantitative magnetic resonance imaging. J Hepatol. 2018 Nov;69(5):1015-1024. doi: 10.1016/j.jhep.2018.05.037. Epub 2018 Jun 8. PMID 29886155
- [Background] Selvaraj EA, Culver EL, Collier J, Ridgway GR, Brady JM, Bailey A, et al. Combination of quantitative MRCP and MRI demonstrates increased periductal iron-corrected T1 in primary sclerosing cholangitis. Gut. 2021;70(Suppl 1):A155.
- [Background] Okada F, Izutsu R, Goto K, Osaki M. Inflammation-Related Carcinogenesis: Lessons from Animal Models to Clinical Aspects. Cancers (Basel). 2021 Feb 22;13(4):921. doi: 10.3390/cancers13040921. PMID 33671768
- [Background] Eaton JE, Talwalkar JA, Lazaridis KN, Gores GJ, Lindor KD. Pathogenesis of primary sclerosing cholangitis and advances in diagnosis and management. Gastroenterology. 2013 Sep;145(3):521-36. doi: 10.1053/j.gastro.2013.06.052. Epub 2013 Jul 1. PMID 23827861
- [Background] Ponsioen CY, Assis DN, Boberg KM, Bowlus CL, Deneau M, Thorburn D, Aabakken L, Farkkila M, Petersen B, Rupp C, Hubscher SG; PSC Study Group. Defining Primary Sclerosing Cholangitis: Results From an International Primary Sclerosing Cholangitis Study Group Consensus Process. Gastroenterology. 2021 Dec;161(6):1764-1775.e5. doi: 10.1053/j.gastro.2021.07.046. Epub 2021 Aug 10. No abstract available. PMID 34384749
- [Background] Luo D, Wan X, Liu J, Tong T. Optimally estimating the sample mean from the sample size, median, mid-range, and/or mid-quartile range. Stat Methods Med Res. 2018 Jun;27(6):1785-1805. doi: 10.1177/0962280216669183. Epub 2016 Sep 27. PMID 27683581
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] McDonald N, Eddowes PJ, Hodson J, Semple SIK, Davies NP, Kelly CJ, Kin S, Phillips M, Herlihy AH, Kendall TJ, Brown RM, Neil DAH, Hubscher SG, Hirschfield GM, Fallowfield JA. Multiparametric magnetic resonance imaging for quantitation of liver disease: a two-centre cross-sectional observational study. Sci Rep. 2018 Jun 15;8(1):9189. doi: 10.1038/s41598-018-27560-5. PMID 29907829
- [Background] Schramm C, Eaton J, Ringe KI, Venkatesh S, Yamamura J; MRI working group of the IPSCSG. Recommendations on the use of magnetic resonance imaging in PSC-A position statement from the International PSC Study Group. Hepatology. 2017 Nov;66(5):1675-1688. doi: 10.1002/hep.29293. Epub 2017 Sep 29. PMID 28555945